CLINICAL TRIAL: NCT01248468
Title: A Multi-center, Randomized, Double-blind, Parallel-group Single-dose, Placebo-controlled Study Comparing the Efficacy and Safety of Acetaminophen, Aspirin and Caffeine With Sumatriptan in the Acute Treatment of Migraine.
Brief Title: Efficacy and Safety of Acetaminophen, Aspirin and Caffeine With Sumatriptan in the Acute Treatment of Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 176-P-401
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-06

CONDITIONS: Pain, Migraine
Keywords: Pain, Migraine
MeSH Terms: conditions — Pain; Migraine Disorders | interventions — acetaminophen, aspirin, caffeine drug combination; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aspirin, acetaminophen and caffeine (Experimental): AAC: 2 tablets, each containing acetaminophen 250 mg, aspiring 250 mg, caffeine 65 mg and 1 placebo tablet matching sumatriptan 100 mg tablets
  Interventions: Drug: Aspirin, acetaminophen and caffeine
- Sumatriptan (100 mg) (Active Comparator): 1 tablet containing sumatriptan 100 mg and 2 placebo tablets matching acetaminophen 250 mg, aspirin 250 mg and caffeine 65 mg tablets
  Interventions: Drug: Sumatriptan
- Placebo (Placebo Comparator): 1 placebo tablet matching sumatriptan 100mg and 2 placebo tablets matching acetaminophen 250 mg, aspirin 250 mg and caffeine 65 mg tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin, acetaminophen and caffeine — 2 tablets each containing Aspirin (250mg), acetaminophen (250mg) and caffeine (65mg)
  Arms: Aspirin, acetaminophen and caffeine
Drug: Sumatriptan — 100 mg Sumatriptan
  Arms: Sumatriptan (100 mg)
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The main purpose of this study is to compare the efficacy and safety of aspirin, acetaminophen and caffeine (AAC) with sumatriptan and placebo in the acute treatment of migraine.

ELIGIBILITY:
Inclusion criteria:

1. Male or female aged 18 years and over.
2. International Headache Society (IHS) diagnosis of migraine without aura or typical aura with migraine headache.
3. History of experiencing at least 1, but not more than 8, acute migraine attacks monthly during the previous year.
4. History of at least moderate migraine pain intensity, if left untreated.

Exclusion criteria:

1. Headache symptoms which may be due to or aggravated by:

   * Recent (within 6 months) head or neck trauma (e.g., whiplash)
   * Head or neck pain secondary to an orthopedic abnormality
   * Cluster headache
   * Specific migraine variants (e.g., basilar-type artery migraine, ophthalmoplegic migraine, hemiplegic migraine, migraine aura without headache)
   * Other serious, non-migraine causes of headache (e.g., increased intracranial pressure, intracranial bleeding, meningitis, malignancy)
   * Non-serious, non-migraine causes of headache (e.g., cold, flu, hangover)
2. Routine use (≥ 10 days per month, on average) of any medication having the potential to interfere with the pharmacologic effects or evaluation of the study medications (e.g., narcotic and non-narcotic analgesic products (prescription or over-the-counter), ergotamine-containing and ergot-type medication, anxiolytics, hypnotics, sedatives, 5HT-1 agonists, anti-emetics, or prokinetic drugs).
3. History of vomiting during more than 20% of migraine episodes or confined to bedrest for more than 50% of migraine episodes.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Leader, Study Director — Novartis Consumer Health
Locations (20):
- United States (20):
  - Anaheim, California
  - San Francisco, California
  - Clearwater, Florida
  - DeLand, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - West Palm Beach, Florida
  - Chicago, Illinois
  - Ann Arbor, Michigan
  - Springfield, Missouri
  - Rochester, New York
  - The Bronx, New York
  - Raleigh, North Carolina
  - Cleveland, Ohio
  - Mt. Pleasant, South Carolina
  - Nashville, Tennessee
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Aspirin, Acetaminophen, and Caffeine: 2 tablets, each containing acetaminophen 250 mg, aspiring 250 mg, caffeine 65 mg and 1 placebo tablet matching sumatriptan 100 mg tablets
Period: Overall Study
Arm/Group | Aspirin, Acetaminophen, and Caffeine | Sumatriptan (100 mg) | Placebo
Started | 299 | 304 | 149
Safety Population | 266 | 271 | 133
ITT Population | 256 | 261 | 125
Completed | 284 | 290 | 145
Not Completed | 15 | 14 | 4
Not completed — Administrative problem | 1 | 0 | 0
Not completed — Lost to Follow-up | 9 | 12 | 4
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin, Acetaminophen, and Caffeine | Sumatriptan (100 mg) | Placebo | Total
Number analyzed (Participants) | 299 | 304 | 149 | 752
Age Continuous [Mean (Standard Deviation); unit: years] | 38 (11.4) | 37.8 (11.4) | 37.6 (11.5) | 37.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250 | 245 | 125 | 620
  Male | 49 | 59 | 24 | 132
Race/Ethnicity, Customized [Number; unit: Participants] — Calculation for randomized subjects
  Participants
    American Indian or Alaska Native | 1 | 1 | 0 | 2
    Asian | 3 | 9 | 5 | 17
    Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
    Black or African American | 44 | 47 | 24 | 115
    White | 244 | 239 | 113 | 596
    Other | 6 | 6 | 7 | 19
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 299 | 304 | 149 | 752

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Who Are Pain Free at 2 Hours.
Description: Subjects assessed severity of pain on a 4 point scale (0=none, …, 3=severe) at set time points after dosing through 4 hours. Subjects who indicated severity of pain=none at 2 hours were considered pain free at 2 hours
Time Frame: 2 hours
Population: The basic population for efficacy analysis was ITT. No explicit process to impute missing values at any given assessment timepoint. Instead, missing values were implicitly imputed by the repeated measures analysis statistical model. So, at any given timepoint, the number of subjects analyzed is slightly less than the total ITT population.
Measure: Number; unit: Percent of participants
Arm/Group | Aspirin, Acetaminophen, and Caffeine | Sumatriptan (100 mg) | Placebo
Number analyzed (Participants) | 248 | 256 | 121
Percent of participants | 34.7 [.938 to 2.484] | 44.9 [0.431 to .900] | 26.4 [1.525 to 3.937]

2. Secondary Outcome: Percent of Subjects Who Are Free of Nausea at 2 Hours.
Description: Subjects assessed severity of relevant symptom on a 4 point scale (0=none, …, 3=severe) at set time points after dosing through 4 hours. Subjects who indicated severity of relevant symptom=none at 2 hours were considered relevant symptom free at 2 hours
Time Frame: 2 hours
Population: The basic population for efficacy analysis was ITT. No explicit process to impute missing values at any given assessment timepoint. Missing values were implicitly imputed by the repeated measures analysis statistical model. Consequently, at any given timepoint, the number of subjects analyzed is slightly less than the total ITT population.
Measure: Number; unit: percent of participants
Arm/Group | Aspirin, Acetaminophen, and Caffeine | Sumatriptan (100 mg) | Placebo
Number analyzed (Participants) | 248 | 252 | 119
percent of participants | 70.6 [.863 to 2.522] | 72.2 [.662 to 1.506] | 66.4 [.856 to 2.549]

3. Secondary Outcome: Percent of Subjects Who Are Free of Phonophobia at 2 Hours.
Description: as for outcome 2
Time Frame: 2 hours
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Aspirin, Acetaminophen, and Caffeine | Sumatriptan (100 mg) | Placebo
Number analyzed (Participants) | 247 | 256 | 119
Percent of participants | 53.4 [.904 to 2.353] | 60.9 [.630 to 1.334] | 46.2 [.977 to 2.590]

4. Secondary Outcome: Percent of Subjects Who Are Free of Photophobia at 2 Hours.
Description: as for outcome 2
Time Frame: 2 hours
Measure: Number; unit: Percent of participants
Arm/Group | Aspirin, Acetaminophen, and Caffeine | Sumatriptan (100 mg) | Placebo
Number analyzed (Participants) | 247 | 256 | 120
Percent of participants | 48.6 [.888 to 2.327] | 52.3 [.631 to 1.315] | 40.8 [.980 to 2.542]

ADVERSE EVENTS:
Arm/Group | Aspirin, Acetaminophen, and Caffeine | Sumatriptan (100 mg) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/266 | 0/271 | 0/133
Other Adverse Events (participants affected / at risk) | 8/266 | 14/271 | 3/133
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aspirin, Acetaminophen, and Caffeine (N=266) | Sumatriptan (100 mg) (N=271) | Placebo (N=133)
Nausea (Gastrointestinal disorders) | 8 | 14 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data of &/or resulting from the performance of the Clinical Trial (CT) shall be pooled with the data from other centers & analyzed as stipulated in the Protocol.Without the consent of the steering committee of the multi-center CT, no presentation/publication of the results obtained from datasets other than the final pooled dataset shall be made prior to the presentation/ publication based on the final pooled dataset.